CLINICAL TRIAL: NCT00005530
Title: Diet, Insulin Resistance, and Cardiovascular Risk
Status: Completed | Type: Observational
Sponsor: University of South Carolina (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5063; R29HL053798 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Insulin Resistance; Hyperinsulinism; Diabetes Mellitus, Non-insulin Dependent; Diabetes Mellitus
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Insulin Resistance; Hyperinsulinism; Diabetes Mellitus, Type 2; Diabetes Mellitus

SUMMARY:
To elucidate dietary factors that elevate risk for cardiovascular disease (CVD) in conjunction with insulin resistance.

DETAILED DESCRIPTION:
BACKGROUND:

Clinical studies indicate that high carbohydrate intake may exacerbate the dyslipidemia often seen with insulin resistance. Consequently, there is much debate as to the optimal dietary pattern for individuals with NIDDM to minimize risk for microvascular disease. Data on this topic from free-living populations are scarce. In addition, associations of dietary antioxidants with CVD risk have not been evaluated in large community samples of persons with diabetes.

DESIGN NARRATIVE:

Potential dietary determinants of hyperinsulinemia or of insulin resistance were evaluated, including high intake of dietary fats and of simple sugars and low alcohol consumption. As a major focus, dietary factors that may contribute to elevated CVD risk among persons with existing insulin resistance, including impaired glucose tolerance (IGT) and non-insulin-dependent diabetes mellitus (NIDDM) were examined. Five datasets from epidemiologic studies were available to evaluate specific hypotheses for men and women of Black, Hispanic and non-Hispanic white ethnicity. The unique contributions of each dataset were as follows. The San Luis Valley Diabetes Study and the San Antonio Heart Study enabled prospective analyses for large numbers of subjects with IGT or NIDDM; the Mexico City Study provided a sample with contrasting dietary patterns in a non-white population; the Kaiser Permanente Women Twins Study allowed for the removal of genetic influences by evaluating associations within monozygotic twin pairs; and the Insulin Resistance Atherosclerosis Study (IRAS) provided direct measurement of insulin sensitivity and subclinical atherosclerosis across the spectrum of glucose tolerance in three ethnic groups.

An understanding of the accuracy of the dietary assessment instruments used in the three ethnic groups was critical to the interpretation of the findings related to diet and CVD risk variables. Therefore, a second component of research was also conducted, that being an evaluation of the comparative validity of the food frequency interview used in the multi- cultural IRAS population using a series of 24-hour dietary recalls as the standard.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-05; Study Completion 2000-04

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Mayer-Davis — University of South Carolina

REFERENCES:
- [Background] Mayer-Davis EJ, Levin S, Marshall JA. Heterogeneity in associations between macronutrient intake and lipoprotein profile in individuals with type 2 diabetes. Diabetes Care. 1999 Oct;22(10):1632-9. doi: 10.2337/diacare.22.10.1632. PMID 10526727
- [Background] Mayer-Davis EJ, Monaco JH, Marshall JA, Rushing J, Juhaeri. Vitamin C intake and cardiovascular disease risk factors in persons with non-insulin-dependent diabetes mellitus. From the Insulin Resistance Atherosclerosis Study and the San Luis Valley Diabetes Study. Prev Med. 1997 May-Jun;26(3):277-83. doi: 10.1006/pmed.1997.0145. PMID 9144749
- [Background] Mayer EJ, Newman B, Austin MA, Zhang D, Quesenberry CP Jr, Edwards K, Selby JV. Genetic and environmental influences on insulin levels and the insulin resistance syndrome: an analysis of women twins. Am J Epidemiol. 1996 Feb 15;143(4):323-32. doi: 10.1093/oxfordjournals.aje.a008746. PMID 8633616
- [Background] Bell RA, Mayer-Davis EJ, Martin MA, D'Agostino RB Jr, Haffner SM. Associations between alcohol consumption and insulin sensitivity and cardiovascular disease risk factors: the Insulin Resistance and Atherosclerosis Study. Diabetes Care. 2000 Nov;23(11):1630-6. doi: 10.2337/diacare.23.11.1630. PMID 11092284